CLINICAL TRIAL: NCT04837430
Title: NT-proBNP and Troponin I in Children With Dengue Hemorrhagic Shock: a Longitudinal Study
Brief Title: NT-proBNP and Troponin I in Dengue Children
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Le Phuoc Truyen (Other)
Responsible Party: Sponsor-Investigator, Le Phuoc Truyen, Clinical Physician, University of Medicine and Pharmacy at Ho Chi Minh City
Organization: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Other Study IDs: 2130-DHYD
Record Dates: First submitted 2021-04-03; First posted 2021-04-08 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Dengue Shock Syndrome; Children, Only
Keywords: NT-proBNP; Troponin I; Dengue children; Cardiac enzyme
MeSH Terms: conditions — Severe Dengue

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To discribe concentration of NT-proBNP and Troponin I in Dengue hemorrhagic shock children, in correlation between concentration of NT-proBNP and troponin I with total fluid admission, respiratory support, using inotrope and vasopressor using.

DETAILED DESCRIPTION:
Treatment of children with Dengue hemorrhagic shock syndrome (DSS) is challenge, especially in cases with hypotensive shock, profound shock or whom do not have a response to initial crystalloid therapy. Currently, treatment of DSS remains almost supportive, with particular emphasis on careful fluid management. However, fluid overload is a common complication of this treatment, lead to many difficulties in management of severe Dengue children, accompany with morbidity and mortality. Diagnosis of fluid overload mostly based on clinical features and chest X-ray or ultrasound. Until now, no biomarker are widely using for diagnosis of fluid overload in clinical. NT-proBNP is secreted when stretching the wall of the cardiac muscle. This may a suitable biomarker to discover the fluid overload state in children with DSS. Troponin I is a biomarker of cardiac muscle damage.

ELIGIBILITY:
Inclusion Criteria:

* Dengue shock children who admitted to ICU

Exclusion Criteria:

* Excluding the cases of children with cardiovascular disease, hyperthyroidism, taking drugs such as insulin, steroid, estrogen, growth hormone, thyroid hormone

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children from 1 month to 15 years old are diagnosed with Dengue shock syndrome according to guidelines of WHO with NS1 (+) or ELISA IgM Dengue (+)
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2021-04-02 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Concentration of NT-proBNP | 10 days
  Concentration of NT-proBNP in Children with Dengue hemorrhagic shock and severe shock
Concentration of Troponin I | 10 days
  Concentration of Troponin I in Children with Dengue hemorrhagic shock and severe shock

SECONDARY OUTCOMES:
Cut-off value of NT-proBNP for fluid overload | 14 days
  Cut-off value of NT-proBNP for pulmonary edema
Correlation between concentration of NT-proBNP | 14 days
  Correlation between concentration of NT-proBNP with total fluid admission, respiratory support, using inotrope and vasopressor using
Correlation between concentration of Troponin I | 14 days
  Correlation between concentration of Troponin I total fluid admission, respiratory support, using inotrope and vasopressor using
Rate of clinical manifestations | 14 days
  Rate of clinical manifestations: fever, abdominal pain, petechia, hematomegaly
Rate of abnormal laboratory exam | 14 days
  electrolyte, arterial blood gas, lactate
Rate of abnormal liver, kidney, hematology laboratory exam | 14 days
  AST, ALT, ure, creatinin, PLT, PT, aPTT, Fibrinogen
Rate of NS1 Dengue | 10 days
  Positive
Rate of MAC ELISA IgM Dengue | 14 days
  Positive
Rate of complications | 14 days
  Pulmonary edema
Rate of respiratory support | 14 days
  Cannula, NCPAP, Intubation
Rate of intubation | 14 days
  Positive
Rate of mode of ventilation | 14 days
  PC, IP, PEEP, FiO2, VT
Total fluid administration | 14 days
  ml/kg/d
Time for IV fluid administration | 14 days
  hours
Rate and kind of cephalosporin using | 14 days
  3rd generation cephalosporin
Rate and kind of Carbapenem using | 14 days
  Carbapenem
Rate and kind of Vancomycin using | 14 days
  Vancomycin
Rate of intraperitoneal fluid drainage | 14 days
  Positive
Rate of CRRT | 14 days
  Positive

CONTACTS AND LOCATIONS:
Overall Officials: Truyen P. Le, MD, Principal Investigator — University of Medicine and Pharmacy at Ho Chi Minh City
Locations (1):
- University of medicine and pharmacy at Ho Chi Minh city, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: No